CLINICAL TRIAL: NCT04684836
Title: Evaluating the Comparative Effectiveness of Telemedicine in Primary Care: Learning From the COVID-19 Pandemic
Brief Title: Comparative Effectiveness of Telemedicine in Primary Care
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20-12023014
Record Dates: First submitted 2020-12-21; First posted 2020-12-28 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease (COPD); Congestive Heart Failure; Diabetes; Hypertension
Keywords: telemedicine; primary care
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Heart Failure; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Telemedicine: Patients in practices that had high telemedicine use, based on the percent of visits the practice delivered via telemedicine from April 2020 to December 2021 (the study post-period)
  Interventions: Other: Exposure to telemedicine, after the onset of the pandemic
- Low Telemedicine: Patients in practices that had some telemedicine use, based on the percent of visits the practice delivered via telemedicine from April 2020 to December 2021 (the study post-period)
  Interventions: Other: Exposure to telemedicine, after the onset of the pandemic

INTERVENTIONS:
Other: Exposure to telemedicine, after the onset of the pandemic — The exposure of interest was the switch to primary care telemedicine prompted by the COVID-19 epidemic

SUMMARY:
Leveraging a natural experiment approach, the investigators will examine rapidly changing telemedicine and in-person models of care during and after the COVID-19 crisis to determine whether certain patients could safely choose to continue telemedicine or telemedicine-supplemented care, rather than return to in-person care.

DETAILED DESCRIPTION:
During the COVID-19 pandemic, telemedicine has quickly emerged as the primary method of providing outpatient care in many regions with shelter-in-place and social distancing policies. It is critical to understand the impact of this rapid and widespread transition from in-person to remote visits on disparities in access to primary care, especially in chronic disease where ongoing communication between providers and patients is essential. Also, these newly developed or expanded telemedicine programs vary widely, raising important questions about the effect of these differences on uptake of telemedicine among different patient populations and on patient-centered outcomes. Leveraging a natural experiment approach, the investigators will examine rapidly changing telemedicine and in-person models of care during and after the COVID-19 crisis to determine whether certain patients could safely choose to continue telemedicine or telemedicine-supplemented care, rather than return to in-person care. The overarching goals of this study are to describe the features of telemedicine programs in primary care during the COVID-19 pandemic and to use natural experiment methods to provide rigorous evidence on the effects of these programs.

PCORI has granted an extension for the final research report to October 1, 2023.

ELIGIBILITY:
Inclusion Criteria:

* patients that are attributed to primary care clinics across four health systems in the INSIGHT (Mount Sinai Health System and Weill Cornell Medicine), OneFlorida (University of Florida Health), and STAR (University of North Carolina Health) CRNs.
* Patients received two or more outpatient visits at a participating practice during a one-year period before the COVID-19 pandemic,
* Patients had one or more of five chronic illnesses (asthma, chronic obstructive pulmonary disease (COPD), congestive heart failure (CHF), diabetes, hypertension) as defined by the Medicare Chronic Conditions Warehouse algorithm

Exclusion Criteria:

* Patients who tested COVID-positive
* Patients from hospice and palliative care practices
* Patients from osteopathic medicine practices
* Patients from pediatric practices
* Patients that did not reside in states where the four health systems were located: the New York-Tri State Area (Connecticut, New York, and New Jersey), Florida, and North Carolina.
* Patients that moved out of state (or out of the New York-Tri State Area) or who died during the study period were also excluded.
* Patients who were not continuously enrolled over the entire study period (2019-2021).

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population encompasses patients that are attributed to primary care clinics in one of the four health systems defined above. Patients are included in the study if they are ages 19 or older and received two or more outpatient visits at a participating practice during a one-year period before the COVID-19 pandemic, and had one or more of five chronic illnesses (asthma, chronic obstructive pulmonary disease (COPD), congestive heart failure (CHF), diabetes, hypertension) as defined by the Medicare Chronic Conditions Warehouse algorithm. For the claims analyses, it will be required that patients are continuously enrolled over the entire study time period.
Sampling Method: Non-Probability Sample
Enrollment: 33100 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Ancker, MPH, PhD, Principal Investigator — Vanderbilt University Medical Center; Rainu Kaushal, MD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - University of Florida, Gainesville, New York
  - Mount Sinai, New York, New York
  - Weill Cornell Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Telemedicine | Low Telemedicine
Started | 17226 | 15874
Completed | 17226 | 15874
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Upon receiving the data from each study site, we first examined the patterns of telehealth provision among all included practices and the extent to which practices could be categorized into one of these three study arms. Given that the data showed an insufficient number of practices would fall into the three original proposed arms, we updated the analytic plan to include two study arms: high- versus low telemedicine practices.
Groups:
- Total: Total of all reporting groups
Arm/Group | High Telemedicine | Low Telemedicine | Total
Number analyzed (Participants) | 17226 | 15874 | 33100
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.64 (10.55) | 71.56 (10.58) | 72.12 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10448 | 9445 | 19893
  Male | 6778 | 6429 | 13207
Race/Ethnicity, Customized [Number; unit: participants]
  White | 12546 | 12489 | 25035
  Black | 5627 | 3030 | 2597
Rural Urban Destination [Count of Participants; unit: Participants]
  Metropolitan | 16195 | 14348 | 30543
  Non-metropolitan | 1031 | 1526 | 2557

OUTCOME MEASURES:

1. Primary Outcome: Preventable Emergency Department (ED) Admissions
Description: Avoidable emergency department (ED) admissions will be obtained from claims data. The Effect of telemedicine on preventable emergency department admissions will be calculated using difference-in-differences methodology. The estimate coefficient of the difference-in-difference model will be reported.
Time Frame: Assessed per person per quarter for 3 years, data collected encompasses retrospective data from Q1 2019 to Q4 2021
Population: Upon receiving the data from each study site, the investigators first examined the patterns of telehealth provision among all included practices and the extent to which practices could be categorized into one of these three study arms. Given that the data showed an insufficient number of practices would fall into the three original proposed arms, the investigators updated the analytic plan to include two study arms: high- versus low telemedicine practices.
Measure: Mean (Inter-Quartile Range); unit: count of ED admissions per person per q
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 17226 | 15874
count of ED admissions per person per q | 0.038 [0 to 0] | 0.048 [0 to 0]
Statistical Analysis 1: Comparison: High Telemedicine vs Low Telemedicine; Test type: Superiority — The analysis leveraged a difference-in-differences research design in an intent-to-treat framework, comparing outcomes for patients receiving care at high-telehealth practices with patients at comparable low-telehealth practices, before relative to after the onset of the pandemic (when telehealth use increased significantly); p = 0.0793, Regression, Linear; All models included practice and year-quarter fixed effects, and clustered standard errors at the practice level; Mean Difference (Net) = -0.0255 — This is the Unadjusted model, which included only an indicator for high telemedicine practice, post-period, and its two-way interaction
Statistical Analysis 2: Comparison: High Telemedicine vs Low Telemedicine; Test type: Superiority — Difference-in-differences model; p = 0.5739, Regression, Linear — This is the fully adjusted regression model, which controlled for patient age group, gender, dual status, race, average percent of 65+ patients, risk score category, rural vs urban, and zip-code level characteristics; Mean Difference (Net) = -0.0786

2. Primary Outcome: Unplanned Hospital Admissions From the ED
Description: Unplanned hospital admissions from the ED will be obtained from claims data. The effect of telemedicine on unplanned hospital admissions will be calculated using difference-in-difference methodology. The estimate coefficient will be reported.
Time Frame: Assessed at the quarter level for 3 years, data collected encompasses retrospective data from Q1 2019 to Q4 2021
Population: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: count of admissions per person per q
Arm/Group | HIgh Telemedicine | Low Telemedicine
Number analyzed (Participants) | 17226 | 15874
count of admissions per person per q | 0.015 [0 to 0] | 0.020 [0 to 0]
Statistical Analysis 1: Comparison: HIgh Telemedicine vs Low Telemedicine; Difference-in-differences model; Test type: Superiority; p = 0.3261, Regression, Linear — This is an adjusted model, which included only an indicator for high telemedicine practice, post-period, and its two-way interaction; Mean Difference (Net) = -0.0014
Statistical Analysis 2: Comparison: HIgh Telemedicine vs Low Telemedicine; Difference-in-differences model; Test type: Superiority; p < 0.01, Regression, Linear — This is a fully adjusted regression model, which controlled for patient age group, gender, dual status, race, average percent of 65+ patients, risk score category, rural vs urban, and zip-code level characteristics; Mean Difference (Net) = 0.0806

3. Primary Outcome: Continuity of Care as Assessed by the Breslau Usual Provider of Care Measure
Description: Continuity of care as assessed by the Breslau Usual Provider of Care measure. The Breslau Usual Provider of Care index is also an indicator of continuity of care, ranging from 0 to 1, where 1 represents continuity of care. The effect of telemedicine on continuity of care using the Breslau Usual Provider of Care measure will be calculated using difference-in-difference methodology. The estimate coefficient will be reported.
Time Frame: Assessed at the quarter level for 3 years, data collected encompasses retrospective data from Q1 2019 to Q4 2021
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: average score on scale by person by q
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 17226 | 15874
average score on scale by person by q | 0.25 [0.14 to 0.50] | 0.35 [0.14 to 0.50]
Statistical Analysis 1: Comparison: High Telemedicine vs Low Telemedicine; Difference-in-differences; Test type: Superiority; p = 0.1101, Regression, Linear — This is an adjusted unadjusted model, which included only an indicator for high telemedicine practice, post-period, and its two-way interaction; Mean Difference (Net) = -0.0217
Statistical Analysis 2: Comparison: High Telemedicine vs Low Telemedicine; Difference-in-differences; Test type: Superiority; p = 0.4618, Regression, Linear — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Net) = 0.5551

4. Primary Outcome: Number of Unplanned Hospital Admissions From the ED
Description: Unplanned hospital admissions from the ED will be obtained from claims data
Time Frame: 60 days after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Continuity of Care as Assessed by the Bice-Boxerman Continuity of Care Index
Description: Continuity of Care as Assessed by the Bice-Boxerman Continuity of Care Index. The Bice-Boxerman Continuity of Care Index is also an indicator of continuity of care, ranging from 0 to 1, where 1 represents continuity of care. The effect of telemedicine on continuity of care using the Bice-Boxerman Continuity of care index will be calculated using difference-in-difference methodology. The estimate coefficient will be reported.
Time Frame: Assessed at the quarter level for 3 years, data collected encompasses retrospective data from Q1 2019 to Q4 2021
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: score on a scale per person per q
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 17226 | 15874
score on a scale per person per q | 0.047 [0.00 to 0.167] | 0.047 [0.00 to 0.0153]
Statistical Analysis 1: Comparison: High Telemedicine vs Low Telemedicine; Difference-in-differences; Test type: Superiority; p = 0.8577, Regression, Linear — This is an unadjusted model, which included only an indicator for high telemedicine practice, post-period, and its two-way interaction; Mean Difference (Net) = -0.0012
Statistical Analysis 2: Comparison: High Telemedicine vs Low Telemedicine; Difference-in-differences; Test type: Superiority; p = 0.5954, Regression, Linear — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Net) = 0.2014

6. Primary Outcome: Number of Unplanned Hospital Admissions From the ED
Description: Unplanned hospital admissions from the ED will be obtained from claims data
Time Frame: 6 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Number of Unplanned Hospital Admissions From the ED
Description: Unplanned hospital admissions from the ED will be obtained from claims data
Time Frame: 12 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Number of Avoidable Emergency Department (ED) Admissions
Description: Avoidable emergency department (ED) admissions will be obtained from claims data
Time Frame: 60 days after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Number of Avoidable Emergency Department (ED) Admissions
Description: Avoidable emergency department (ED) admissions will be obtained from claims data
Time Frame: 6 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Number of Avoidable Emergency Department (ED) Admissions
Description: Avoidable emergency department (ED) admissions will be obtained from claims data
Time Frame: 12 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Continuity of Care as Assessed by the Bice-Boxerman Continuity of Care Index
Description: Continuity of care will be measured using the Bice-Boxerman Continuity of Care Index. The Bice-Boxerman continuity of care (COC) index reflects the relative share of all of a patient's visits during the year that are billed by distinct providers and/or practices. The index ranges from 0 to 1, where 0 indicates that each visit involved a different provider than all other visits, and 1 that all visits were billed by a single provider, representing continuity of care.
Time Frame: 60 days after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Continuity of Care as Assessed by the Bice-Boxerman Continuity of Care Index
Description: as for outcome 11
Time Frame: 6 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Continuity of Care as Assessed by the Bice-Boxerman Continuity of Care Index
Description: as for outcome 11
Time Frame: 12 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Continuity of Care as Assessed by the Breslau Usual Provider of Care Measure
Description: Continuity of care as assessed by the Breslau Usual Provider of Care measure. The Breslau Usual Provider of Care index is also an indicator of continuity of care, ranging from 0 to 1, where 1 represents continuity of care.
Time Frame: 60 days after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Continuity of Care as Assessed by the Breslau Usual Provider of Care Measure
Description: as for outcome 14
Time Frame: 6 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

16. Primary Outcome: Continuity of Care as Assessed by the Breslau Usual Provider of Care Measure
Description: as for outcome 14
Time Frame: 12 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

17. Primary Outcome: Continuity of Care as Assessed by Attendance at Follow-up Appointment
Description: Continuity of care as assessed by attendance at follow-up appointment.
Time Frame: 30 days after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

18. Primary Outcome: Continuity of Care as Assessed by Attendance at Follow-up Appointment
Description: Continuity of care as assessed by attendance at follow-up appointment.
Time Frame: 60 days after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

19. Primary Outcome: Continuity of Care as Assessed by Attendance at Follow-up Appointment
Description: Continuity of care as assessed by attendance at follow-up appointment.
Time Frame: 6 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

20. Primary Outcome: Continuity of Care as Assessed by Attendance at Follow-up Appointment
Description: Continuity of care as assessed by attendance at follow-up appointment.
Time Frame: 12 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Evidence of Controlled Disease as Indicated by as Indicated by the National Quality Forum (NQF 0059): Diabetes: Hemoglobin A1c (HbA1c) Poor Control (>9%)
Description: Evidence of controlled disease as indicated by as indicated by the National Quality Forum (NQF 0059): Diabetes: Hemoglobin A1c (HbA1c) Poor Control (>9%), which is the percentage of patients 18 - 75 years of age with diabetes who had hemoglobin A1c > 9.0% during the measurement period
Time Frame: 30 days after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Evidence of Controlled Disease as Indicated by as Indicated by the National Quality Forum (NQF 0059): Diabetes: Hemoglobin A1c (HbA1c) Poor Control (>9%)
Description: as for outcome 21
Time Frame: 60 days after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Evidence of Controlled Disease as Indicated by as Indicated by the National Quality Forum (NQF 0059): Diabetes: Hemoglobin A1c (HbA1c) Poor Control (>9%)
Description: as for outcome 21
Time Frame: 6 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Evidence of Controlled Disease as Indicated by as Indicated by the National Quality Forum (NQF 0059): Diabetes: Hemoglobin A1c (HbA1c) Poor Control (>9%)
Description: as for outcome 21
Time Frame: 12 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Evidence of Controlled Disease as Indicated by as Indicated by the National Quality Forum (NQF 0018): Controlling High Blood Pressure
Description: Evidence of controlled disease as indicated by as indicated by the National Quality Forum (NQF 0018): Controlling High Blood Pressure, which is the percentage of patients 18 - 85 with hypertension diagnosis and adequate control (< 140/90 mmHg)
Time Frame: 30 days after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Evidence of Controlled Disease as Indicated by as Indicated by the National Quality Forum (NQF 0018): Controlling High Blood Pressure
Description: as for outcome 25
Time Frame: 60 days after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Evidence of Controlled Disease as Indicated by as Indicated by the National Quality Forum (NQF 0018): Controlling High Blood Pressure
Description: as for outcome 25
Time Frame: 6 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Evidence of Controlled Disease as Indicated by as Indicated by the National Quality Forum (NQF 0018): Controlling High Blood Pressure
Description: as for outcome 25
Time Frame: 12 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Days at Home
Description: Days per month not in hospital or institutional setting
Time Frame: 30 days after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Days at Home
Description: Days per month not in hospital or institutional setting
Time Frame: 60 days after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Days at Home
Description: Days per month not in hospital or institutional setting
Time Frame: 6 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Days at Home
Description: Days per month not in hospital or institutional setting
Time Frame: 12 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Patient Experiences Based on the Patient Satisfaction Questionnaire (PSQ-18)
Description: Patient experiences based on the Patient Satisfaction Questionnaire (PSQ-18), which is a 5-scale questionnaire including questions on patient satisfaction, communication quality with providers and accessibility/convenience of care.
Time Frame: 12 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Ease of Use and Access to Telemedicine Based on Telehealth Usability Questionnaire (TUQ)
Description: For individuals who accessed a telemedicine visit, we will ask questions based on the validated Telehealth Usability Questionnaire (TUQ), including the ease of use and access to the telemedicine service, quality of the interaction with the provider, and satisfaction
Time Frame: 12 months after the exposure to one of the comparator arms of clinic-level telemedicine used
Population: Data was not collected for this measure.
Arm/Group | High Telemedicine | Low Telemedicine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected.
Description: Adverse event data were not collected.
Arm/Group | HIgh Telemedicine | Low Telemedicine
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT04684836/Prot_SAP_000.pdf